CLINICAL TRIAL: NCT01135017
Title: A Placebo-Controlled, Double-Blind, Randomized, Multi-Center Study to Assess the Effects of Dronedarone 400 mg BID for 12 Weeks on Atrial Fibrillation Burden in Subjects With Permanent Pacemakers
Brief Title: Effects of Dronedarone on Atrial Fibrillation Burden in Subjects With Permanent Pacemakers
Acronym: HESTIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRONE_L_04316; U1111-1117-0024 (Other: UTN)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2013-04-01 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone (Experimental): Dronedarone 400 mg twice a day for 12 weeks
  Interventions: Drug: Dronedarone
- Placebo (Placebo Comparator): Placebo (for Dronedarone) twice a day for 12 weeks
  Interventions: Drug: Placebo (for Dronedarone)

INTERVENTIONS:
Drug: Dronedarone — Film-coated tablet
  Oral administration under fed conditions (during breakfast and dinner)
  Other Names: Multaq®; SR33589
  Arms: Dronedarone
Drug: Placebo (for Dronedarone) — Film-coated tablet strictly identical in appearance
  Oral administration under fed conditions (during breakfast and dinner)
  Arms: Placebo

SUMMARY:
Primary objective was to evaluate the effects of dronedarone on Atrial Fibrillation (AF) burden (i.e. percent time in AF) as measured on electrogram (EGM) in subjects with a permanent pacemaker.

Secondary objectives were to evaluate:

* the effects of dronedarone on AF pattern characteristics i.e. ventricular rate during AF;
* the effects of dronedarone on subject-perceived AF burden and symptom severity as reported by subjects using the Atrial Fibrillation Severity Scale (AFSS);
* the incidence of electrical cardioversion (or overdrive pacing) during treatment;
* the safety of dronedarone.

DETAILED DESCRIPTION:
The maximum duration of the study period for a participant was 18 weeks (approximatively 4.5 months) including up to 4 weeks screening, 12-week Treatment period and a post-treatment follow-up of 2 weeks.

ELIGIBILITY:
Inclusion criteria:

* Paroxysmal AF or atrial flutter (AFL) documented by evidence of AF/AFL and sinus rhythm within the prior 6 months;
* AF burden ≥1% on pacemaker EGM interrogation at screening, with at least one episode of AF within the previous 28 days;
* Programmable dual chamber pacemaker with lead placement no less than 3 months before screening, a minimum capability of storing 3 months or more of EGM data, and an expected remaining battery life of 1 year or more.

Exclusion criteria:

* AF burden <1% on pacemaker EGM interrogation at screening;
* None of the following cardiovascular risk factors: Age ≥70 years, hypertension, diabetes mellitus, prior cardiovascular accident or systemic embolism, left atrium diameter ≥50 mm by M-mode or 2D echocardiography, or left ventricular ejection fraction ≤0.40 by M-mode or 2D echocardiography, cardiac catheterization, or nuclear cardiac imaging;
* Permanent AF;
* Evidence of persistent AF (continuous AF activity lasting longer than 7 days);
* Electrical cardioversion (or overdrive pacing) within 4 weeks prior to screening;
* Cardiac ablation procedure within 3 months prior to screening;
* Evidence of uncorrected atrial undersensing or oversensing documented in routine pacemaker evaluation at screening;
* Pacemaker programming requirements for the study not clinically feasible, contraindicated, or could have posed risk;
* Ongoing potentially dangerous symptoms when in AF/AFL such as angina pectoris, transient ischemic attacks, stroke, or syncope;
* New York Heart Association (NYHA) Class IV heart failure or NYHA Class II or III heart failure with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic within 4 weeks prior to screening;
* Evidence of clinical instability including hypotension, unstable angina and hemodynamically significant obstructive valvular disease, hemodynamically significant obstructive cardiomyopathy, a cardiac operation, or revascularization procedure within 4 weeks prior to screening;
* Noncardiovascular illness or disorder that could have precluded participation or severely limit survival including cancer with metastasis and organ transplantation requiring immune suppression;
* Planned noncardiac or cardiac surgery or procedures including surgery for valvular heart disease, coronary artery bypass graft, percutaneous coronary intervention, cardiac transplantation or electrical cardioversion for AF/AFL;
* Need for concomitant medication that were prohibited in this trial: Antiarrhythmics, drugs or products that are strong inhibitors of CYP3A, CYP3A inducers;
* Chronic use of amiodarone within the 4 weeks prior to screening;
* Use of Class I or Class III antiarrhythmics (other than amiodarone) within 5-half lives prior to screening;
* Use of St John's wort, grapefruit juice, or drugs that prolong the QT interval and might have increased the risk of torsade de pointes;
* Inability or unwillingness to comply with oral anticoagulation therapy, if indicated;
* Bazett corrected QT interval interval ≥500 msec at screening (if in sinus rhythm);
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥ 100mmHg) at screening;
* Uncorrected hypokalemia (serum potassium <3.5 mEq/L)
* Severe hepatic impairment (ie, Child-Pugh Class C), abnormal liver function test defined as alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin >2 X upper limit of normal (ULN), or renal impairment defined as serum creatinine >2.0 mg/dL at screening;
* Uncontrolled diabetes mellitus (documented history of HbA1c >10% at the most recent assessment prior to screening);
* Pregnant woman or woman of childbearing potential not on adequate birth control;
* Breastfeeding woman;
* Previous (within 2 months prior to screening) or current participation in another clinical trial with an investigational drug (under development) or investigational device.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (92):
- United States (92):
  - Investigational Site Number 840015, Birmingham, Alabama
  - Investigational Site Number 840087, Huntsville, Alabama
  - Investigational Site Number 840018, Mobile, Alabama
  - Investigational Site Number 840030, Mesa, Arizona
  - Investigational Site Number 840048, Phoenix, Arizona
  - Investigational Site Number 840072, Phoenix, Arizona
  - Investigational Site Number 840013, Tucson, Arizona
  - Investigational Site Number 840069, Hot Springs, Arkansas
  - Investigational Site Number 840121, Beverly Hills, California
  - Investigational Site Number 840090, Laguna Hills, California
  - Investigational Site Number 840068, Los Angeles, California
  - Investigational Site Number 840062, Mission Hills, California
  - Investigational Site Number 840070, Orange, California
  - Investigational Site Number 840021, Riverside, California
  - Investigational Site Number 840024, San Diego, California
  - Investigational Site Number 840001, Aurora, Colorado
  - Investigational Site Number 840089, Littleton, Colorado
  - Investigational Site Number 840029, Loveland, Colorado
  - Investigational Site Number 840108, Newark, Delaware
  - Investigational Site Number 840045, Washington D.C., District of Columbia
  - Investigational Site Number 840106, Washington D.C., District of Columbia
  - Investigational Site Number 840010, Clearwater, Florida
  - Investigational Site Number 840020, Fort Myers, Florida
  - Investigational Site Number 840058, Inverness, Florida
  - Investigational Site Number 840043, Jacksonville, Florida
  - Investigational Site Number 840066, Jacksonville, Florida
  - Investigational Site Number 840128, Jacksonville, Florida
  - Investigational Site Number 840044, Jacksonville Beach, Florida
  - Investigational Site Number 840042, Orlando, Florida
  - Investigational Site Number 840016, Port Charlotte, Florida
  - Investigational Site Number 840080, Wellington, Florida
  - Investigational Site Number 840056, Gainesville, Georgia
  - Investigational Site Number 840092, Normal, Illinois
  - Investigational Site Number 840032, Oak Lawn, Illinois
  - Investigational Site Number 840046, Rockford, Illinois
  - Investigational Site Number 840051, Bloomington, Indiana
  - Investigational Site Number 840053, Kansas City, Kansas
  - Investigational Site Number 840110, Owensboro, Kentucky
  - Investigational Site Number 840102, Columbia, Maryland
  - Investigational Site Number 840017, Lansing, Michigan
  - Investigational Site Number 840081, Lapeer, Michigan
  - Investigational Site Number 840075, Petoskey, Michigan
  - Investigational Site Number 840027, Troy, Michigan
  - Investigational Site Number 840104, Saint Cloud, Minnesota
  - Investigational Site Number 840097, Tupelo, Mississippi
  - Investigational Site Number 840037, Columbia, Missouri
  - Investigational Site Number 840035, Kansas City, Missouri
  - Investigational Site Number 840060, St Louis, Missouri
  - Investigational Site Number 840055, St Louis, Missouri
  - Investigational Site Number 840067, Missoula, Montana
  - Investigational Site Number 840049, Reno, Nevada
  - Investigational Site Number 840054, Reno, Nevada
  - Investigational Site Number 840026, Bridgewater, New Jersey
  - Investigational Site Number 840093, Englewood, New Jersey
  - Investigational Site Number 840006, Buffalo, New York
  - Investigational Site Number 840077, Kingston, New York
  - Investigational Site Number 840096, Mineola, New York
  - Investigational Site Number 840041, Syracuse, New York
  - Investigational Site Number 840036, The Bronx, New York
  - Investigational Site Number 840086, Troy, New York
  - Investigational Site Number 840007, Williamsville, New York
  - Investigational Site Number 840084, Raleigh, North Carolina
  - Investigational Site Number 840061, Wilmington, North Carolina
  - Investigational Site Number 840065, Tulsa, Oklahoma
  - Investigational Site Number 840008, Camp Hill, Pennsylvania
  - Investigational Site Number 840009, Doylestown, Pennsylvania
  - Investigational Site Number 840004, Philadelphia, Pennsylvania
  - Investigational Site Number 840078, Phoenixville, Pennsylvania
  - Investigational Site Number 840105, Pittsburgh, Pennsylvania
  - Investigational Site Number 840130, Scranton, Pennsylvania
  - Investigational Site Number 840019, Unionville, Pennsylvania
  - Investigational Site Number 840023, Wyomissing, Pennsylvania
  - Investigational Site Number 840119, Greenville, South Carolina
  - Investigational Site Number 840002, Rapid City, South Dakota
  - Investigational Site Number 840114, Germantown, Tennessee
  - Investigational Site Number 840118, Corpus Christi, Texas
  - Investigational Site Number 840014, Dallas, Texas
  - Investigational Site Number 840012, San Antonio, Texas
  - Investigational Site Number 840125, Tyler, Texas
  - Investigational Site Number 840083, Salt Lake City, Utah
  - Investigational Site Number 840113, Danville, Virginia
  - Investigational Site Number 840082, Lynchburg, Virginia
  - Investigational Site Number 840088, Manassas, Virginia
  - Investigational Site Number 840099, Richmond, Virginia
  - Investigational Site Number 840112, Richmond, Virginia
  - Investigational Site Number 840003, Tacoma, Washington
  - Investigational Site Number 840107, Tacoma, Washington
  - Investigational Site Number 840123, Green Bay, Wisconsin
  - Investigational Site Number 840022, Madison, Wisconsin
  - Investigational Site Number 840033, Milwaukee, Wisconsin
  - Investigational Site Number 840047, Milwaukee, Wisconsin
  - Investigational Site Number 840076, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated in July 2010 was discontinued in December, 2011 due to significantly lower than planned enrollment with no feasibility to complete the trial within reasonable, meaningful timelines and despite a protocol amendment that extended the recruitment period and reduced the sample size from 424 to 286 participants.
Pre-assignment Details: After signature of the informed consent and after eligibility was confirmed, group assignment was made at site in a 1:1 ratio using a treatment code list generated centrally by Sanofi. Participants were considered as randomized as soon as the assignment was made.
  Only 112 patients were randomized at 62 sites.
Period: Overall Study
Arm/Group | Placebo | Dronedarone
Started | 55 | 57
Treated | 55 | 57
Evaluable for Efficacy | 55 | 55 (Two participants did not have interrogation of the pacemaker after randomization)
Completed | 49 (The study was terminated after enrolled participants completed the study period as per protocol) | 45 (The study was terminated after enrolled participants completed the study period as per protocol)
Not Completed | 6 | 12
Not completed — Adverse Event | 3 | 8
Not completed — Other than above | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dronedarone | Total
Number analyzed (Participants) | 55 | 57 | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 74.5 (9.5) | 77.3 (8.6) | 75.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 28 | 45
  Male | 38 | 29 | 67

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation (AF) Burden During the 12-week Treatment Period
Description: AF burden, defined as the percent time a subject is in AF, was evaluated centrally by a Pacemaker Core Lab based on pacemaker interrogation reports including Electrogram (EGM) data provided by the Investigator.
  AF burden during the 12-week treatment period was defined as the duration-weighted average of AF burden collected at Week 4 and Week 12. It was calculated from the single available measurement when one measurement was missing.
Time Frame: Baseline (before randomization), 4 weeks and 12 weeks after randomization
Population: The analysis included all randomized and treated participants with post-baseline AF burden assessment. Participants were included in the treatment group to which they were randomized (Modified Intent-to-treat analysis).
Measure: Geometric Mean (95% Confidence Interval); unit: percent time in AF
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 55 | 55
percent time in AF
  Baseline | 8.77 [6.413 to 12.006] | 10.14 [7.167 to 14.354]
  12-week treatment period | 9.90 [6.633 to 14.772] | 4.63 [2.610 to 8.198]
Statistical Analysis 1: Comparison: Placebo vs Dronedarone; The planned sample size of 286 participants was estimated to have 70% power to detect a reduction in mean AF burden of 30% relative to the placebo group. Due to the smaller-than-planned sample size, the power to detect this difference was estimated to be only 44%, based on the original assumption. However, the power to detect larger treatment effects (>40% reduction) remained high and the posthoc power to detect a 60% reduction in AF burden was 99%; Test type: Superiority or Other; p = 0.0015, ANCOVA — No adjustment for multiplicity was made. The priori threshold for statistical significance was ≤0.05; ANCOVA model on log-transformed AF burden data with treatment arm as a fixed effect term and baseline log-transformed AF burden as a covariate; Least Squares (LS) Mean difference = -59.13, 95% CI 2-sided [-76.322 to -29.457], Standard Error of Mean 0.275 — Percent change in AF burden with dronedarone relative to placebo LS Mean difference from the ANCOVA model on log-transformed AF burden data was exponentiated to convert back to percent change

2. Secondary Outcome: AF Burden During the First 4 Weeks of Treatment and After 4-week Treatment
Description: AF burden at each pacemaker interrogation as evaluated centrally by the Pacemaker Core Lab
Time Frame: 4 weeks and 12 weeks after randomization
Population: Modified intent-to-treat population as previously defined
Measure: Geometric Mean (95% Confidence Interval); unit: percent time in AF
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 55 | 55
percent time in AF
  Week 1 - 4 (n =54, 49) | 8.99 [5.901 to 13.705] | 3.62 [1.806 to 7.258]
  Week 5 - 12 (n =54, 54) | 9.37 [5.938 to 14.786] | 4.28 [2.388 to 7.673]

3. Secondary Outcome: Average Ventricular Rate During AF Episodes
Description: Ventricular rates of AF episodes were obtained from pacemaker interrogation and EGM review.
  The average ventricular rate during AF episodes in the 12-week treatment period was defined as the duration-weighted average of the ventricular rates collected at Week 4 and Week 12. It was calculated from the single available measurement when one measurement was missing.
Time Frame: Baseline (before randomization), 4 weeks and 12 weeks after randomization
Population: Modified intent-to-treat population as previously defined
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 55 | 55
beats/min
  Baseline (n =49, 47) | 93.02 (16.74) | 90.68 (19.80)
  Week 1-12 (n =49, 48) | 95.67 (17.43) | 91.28 (20.30)
  --- Week 1-4 (n =44, 41) | 96.80 (20.09) | 91.93 (21.89)
  --- Week 5-12 (n =47, 42) | 95.58 (18.72) | 88.56 (20.69)

4. Secondary Outcome: Atrial Fibrillation Severity Scale (AFSS) Scores
Description: The University of Toronto Atrial Fibrillation Severity Scale is an instrument to assess the subject-perceived AF burden and AF symptom severity. It consists in a questionnaire plus a scoring algorithm.
  AF Burden score ranges from 3 to 30 and higher scores indicate greater AF burden.
  AF symptoms severity score ranges from 0 to 35 and higher scores indicate extremely severe AF symptoms.
Time Frame: Baseline (before randomization) and 12 weeks after randomization
Population: Modified intent-to-treat population as previously defined
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 55 | 55
units on a scale
  AF burden at baseline (n =45, 34) | 13.72 (4.59) | 12.76 (4.62)
  AF burden after 12-week treatment (n =38, 31) | 13.30 (5.40) | 12.48 (5.45)
  AF symptoms at baseline (n =55, 55) | 8.47 (6.97) | 8.36 (6.83)
  AF symptoms after 12-week treatment (n =54, 53) | 8.06 (7.11) | 7.42 (7.48)

5. Secondary Outcome: Incidence Rate of Electrical Cardioversion (or Overdrive Pacing)
Description: Electrical cardioversion is a procedure in which an electric shock is used to restore normal heart rhythm. Overdrive pacing is a procedure in which an artificial cardiac pacemaker is used to increase the heart rate in order to suppress certain arrhythmias.
  Incidence rate of electrical cardioversion (or overdrive pacing) is expressed as the number of participants that was cardioverted or paced during the study.
Time Frame: 12 weeks
Population: Modified intent-to-treat population as previously defined
Measure: Number; unit: participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 55 | 55
participants | 1 | 0

6. Other Pre Specified Outcome: Overview of Adverse Events (AE)
Description: AE are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: from first study drug intake up to 10 days after the last study drug intake
Population: All randomized and treated participants. Participants were considered according to the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 55 | 57
participants
  Any AE | 31 | 37
  - Any serious AE | 7 | 7
  - Any AE leading to death | 0 | 0
  - Any AE leading to treatment discontinuation | 3 | 8

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected regardless of seriousness or relationship to the drug in the period spanning from signature of the Informed Consent Form up to the last visit.
Description: The analysis included all randomized participants who received at least one dose of study drug and all AE that developed or worsened from randomization up to 10 days after last study drug intake.
  Participants were considered according to the treatment actually received regardless the amount of treatment administered.
Arm/Group | Placebo | Dronedarone
Serious Adverse Events (participants affected / at risk) | 7/55 | 7/57
Other Adverse Events (participants affected / at risk) | 9/55 | 16/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Dronedarone (N=57)
Lobar pneumonia (Infections and infestations) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardiomyopathy (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Dronedarone (N=57)
Dizziness (Nervous system disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 1 | 7
Fatigue (General disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Due to smaller-than-planned number of participants (112 instead of 424), results should be cautiously interpreted. However, the power to detect large treatment effect remained high and the posthoc power to detect a 60% reduction in AF burden was 99%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can present or publish trial results. A copy is submitted to the Sponsor for review and comment at least 45 days in advance of the submission to journal (20 days for abstracts).

The Sponsor can require to delay the communication for a period not exceeding 90 days to allow for filing a patent application or such other measures as Sponsor deems appropriate to establish and preserve its proprietary rights.